CLINICAL TRIAL: NCT03758482
Title: Factors That Determine the Responses to Meal Ingestion: Effect of Gender on Sensory and Metabolomic Responses
Brief Title: Biological Response to Meal Ingestion: Gender Differences
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PR(AG)338/2016F
Record Dates: First submitted 2018-11-16; First posted 2018-11-29 (Actual); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Healthy
Keywords: meal ingestion; metabolomic responses; hedonic sensations; homeostatic sensations

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Men (Other): The probe meal consists of: 50 g fatty liver duck, 15 g toasts, 50 g cheese, 25 g potato chips, 10 g salted peanuts and 140 mL soft drink.
  Interventions: Other: Probe meal
- Women (Other): The probe meal consists of: 50 g fatty liver duck, 15 g toasts, 50 g cheese, 25 g potato chips, 10 g salted peanuts and 140 mL soft drink.
  Interventions: Other: Probe meal

INTERVENTIONS:
Other: Probe meal — The probe meal (total caloric content 750 Kcal) will be ingested at a standard rate in 10 min.

SUMMARY:
Aim: to determine the effect of gender on the sensory and metabolomic responses to a standard probe meal. Participants (12 men and 12 women) will be instructed to eat a standard dinner the day before, to consume a standard breakfast at home after overnight fast, and to report to the laboratory, where the test meal will be administered 4 h after breakfast. Studies will be conducted in a quiet, isolated room with participants sitting on a chair. Participants will ingest a standard probe meal (750 Kcal). Perception of homeostatic sensations (hunger/satiation, fullness) and hedonic sensations (digestive well-being, mood) will be measured at 5 min intervals 10 min before and 20 min after ingestion and at 10 min intervals up to 60 min after the probe meal. Heart rate variability, blood pressure and body temperature were measured before and after the meal. Blood samples for metabolomic analysis were taken before and 30 min after the meal.

ELIGIBILITY:
Inclusion Criteria:

* Non obese

Exclusion Criteria:

* history of gastrointestinal symptoms
* prior obesity
* use of medications
* history of anosmia and ageusia
* current dieting
* alcohol abuse
* psychological disorders
* eating disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-11-16 (Actual)

PRIMARY OUTCOMES:
Fullness sensation induced by the probe meal | 1 day
  Gender differences in fullness sensation [(measured by a 10 cm scale graded from 0 (not at all) to 10 (very much)] by repeated measures ANCOVA (dependent variable: postprandial sensations scores; between and within subject's factors: gender and time, respectively; covariate: premeal scores).

SECONDARY OUTCOMES:
Change in hunger/satiety induced by the probe meal | 1 day
  Gender differences in hunger/satiety [(measured by a 10 cm scale graded from -5 (extremely hungry) to +5 (completely satiate)] by repeated measures ANCOVA (dependent variable: postprandial sensations scores; between and within subject's factors: gender and time, respectively; covariate: premeal scores).
Change in digestive well-being induced by the probe meal | 1 day
  Gender differences in digestive well-being [(measured by a 10 cm scale graded from -5 (extremely unpleasant sensation) to +5 (extremely pleasant sensation)] by repeated measures ANCOVA (dependent variable: postprandial sensations scores; between and within subject's factors: gender and time, respectively; covariate: premeal scores).
Change in mood induced by the probe meal | 1 day
  Gender differences in mood [(measured by a 10 cm scale graded from -5 (negative) to +5 (postive)] by repeated measures ANCOVA (dependent variable: postprandial sensations scores; between and within subject's factors: gender and time, respectively; covariate: premeal scores).
Change in circulating metabolites induced by the probe meal | 1 day
  Change in low-molecular weight metabolites and lipoproteins analysed using nuclear magnetic resonance.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Result] Pribic T, Azpiroz F. Biogastronomy: Factors that determine the biological response to meal ingestion. Neurogastroenterol Motil. 2018 Jul;30(7):e13309. doi: 10.1111/nmo.13309. Epub 2018 Feb 2. PMID 29392797